CLINICAL TRIAL: NCT00150241
Title: A Seven-Week Double-Blind, Placebo-Controlled, Randomized, Multicenter Study Evaluating the Safety and Efficacy of Three Doses of CP-526,555 ( 0.3 mg QD, 1 mg QD, and 1 mg BID ) in Comparison With Zyban in Smoking Cessation
Brief Title: A Seven-Week Dose-Ranging Study of CP-526,555 Compared With Placebo and Zyban for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051002
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

INTERVENTIONS:
Drug: CP-526,555 (varenicline)

SUMMARY:
The purpose of the study is to measure the safety and efficacy of three doses of varenicline for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have smoked on average of at least ten cigarettes per day during the past year
* Subjects must have no period of abstinence greater than three months in the past year

Exclusion Criteria:

* Subjects with any history of cardiovascular disease
* Myocardial infarction
* Significant arrhythmias
* Poorly controlled hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625
Dates: Start 2000-02; Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome is smoking abstinence for any continuous 4-week period (4-week CQR) during the study treatment phase.

SECONDARY OUTCOMES:
Fixed window 4-week CQR, Weeks 3-6, 4-7
Continuous abstinence from Target Quit Date to Weeks 12, 24, and 52
7-day Point Prevalence of abstinence Week 52
Number of cigarettes smoked per day
Minnesota Nicotine Withdrawal Scale
Smoking Effects Inventory
Brief Questionnaire of Smoking Urge

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Morgantown, West Virginia

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051002